CLINICAL TRIAL: NCT00050167
Title: Evaluation of Differing Taxanes/Taxane Combinations on the Outcome of Patients With Operable Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID01-580
Record Dates: First submitted 2002-11-25; First posted 2002-11-27 (Estimated); Results first posted 2011-08-05 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2011-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Capecitabine; Docetaxel; Paclitaxel; Taxotere; Taxol; Xeloda; Taxanes; Operable Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Docetaxel; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Weekly Paclitaxel (WP) (Experimental): Weekly Paclitaxel (WP) for 12 weeks followed by Fluorouracil + Epirubicin + Cyclophosphamide (FEC) every 3 weeks for 4 cycles
  Interventions: Drug: Paclitaxel
- Docetaxel and Capecitabine (DX) (Experimental): Docetaxel + Capecitabine (DX) days 1-14 every 3 weeks for 4 cycles followed by FEC for 4 cycles.
  Interventions: Drug: Docetaxel; Drug: Capecitabine

INTERVENTIONS:
Drug: Paclitaxel — 80 mg/m^2 by vein (IV) Weekly Over 1 Hour x 12 Weeks
  Other Names: Taxol
  Arms: Weekly Paclitaxel (WP)
Drug: Docetaxel — 75 mg/m^2 by vein (IV) Over 1 Hour Once Every 3 Weeks
  Other Names: Taxotere
  Arms: Docetaxel and Capecitabine (DX)
Drug: Capecitabine — 1500 mg/m^2 by mouth Twice Daily x 2 Weeks
  Other Names: Xeloda
  Arms: Docetaxel and Capecitabine (DX)

SUMMARY:
Primary Objectives:

* Determine the impact of each regimen on the disease free and overall survival of patients with operable breast cancer.
* Determine the ability of docetaxel/capecitabine to downstage primary breast cancer when administered in the neoadjuvant setting when compared with weekly paclitaxel.
* Determine the ability of each regimen to enhance breast conservation therapy when administered in the neoadjuvant setting. (See protocol text for additional objectives and details).

DETAILED DESCRIPTION:
Before the study, participants will have a complete physical exam, including blood tests and a chest x-ray. A mammogram and a sonogram of the breast and armpit will be done to record tumor size (for patients who have not had surgery). Sonography of the liver or a CT scan of the abdomen will also be done. In some patients who have not had surgery, 3-4 samples of the breast tumor will be taken to help confirm the diagnosis of breast cancer. A biopsy needle will be used to collect the samples.

During the study, participants will have blood tests done before each dose of chemotherapy. For participants who have not had surgery, a mammogram and sonogram will be done of the breast and armpit after completion of paclitaxel or docetaxel/capecitabine and after completion of fluorouracil, cyclophosphamide, and epirubicin (FEC). These studies will help doctors to keep track of the tumor size and help with the final decision whether to remove all or part of the breast and nearby lymph nodes after completion of chemotherapy.

Participants in this study will be randomly assigned (as in the toss of a coin) to one of two treatment groups. There is an equal chance of being in either group.

Participants in Group I will receive paclitaxel once a week. The drug will be given through a plastic tube in a vein over 1 hour for a total of 12 treatments. Before each treatment, patients will receive the drug Decadron (dexamethasone) through the vein and may receive Zofran (ondansetron), Benadryl (diphenhydramine hydrochloride) and/or cimetidine to help decrease the risk of side effects from paclitaxel.

Participants in Group II will receive docetaxel and capecitabine. Docetaxel will be given once every 3 weeks. Docetaxel will be given through a plastic tube in the vein over 1 hour. Capecitabine will be started the same day docetaxel is given. This medicine is given in a pill form. The doctor will prescribe a dose of these pills based upon body weight and height. Participants will take several pills two times a day for 14 days. Participants will then not take any capecitabine pills for one week, until the next dose of docetaxel is given. This combination of docetaxel and capecitabine will be given four times (over a period of 12 weeks). Before each treatment, patients will receive the drug Decadron (dexamethasone) by mouth.

After treatment with either paclitaxel or docetaxel/capecitabine, all participants will receive the drugs FEC through a plastic tube into a vein. All of these drugs will be given once every three weeks for a total of 4 treatments (12 weeks total). Decadron (dexamethasone), Zofran (ondansetron) and Benadryl (diphenhydramine hydrochloride) will be given before the chemotherapy to help decrease the risk of side effects.

Participants who have a Her-2/neu positive cancer will potentially be eligible to receive trastuzumab therapy for 1 year. This medicine is given through a vein either once a week (over 30 minutes) or once every 3 weeks (over 30 minutes). Your doctor will discuss whether this medicine is appropriate for you.

After all treatment is done, participants whose tumors are sensitive to hormones (estrogen) will take a pill to help decrease the amount of hormone (estrogen) that can reach any tumor cells. This pill will be taken once a day for 5 years.

Participants who have not completed surgery for their cancer before receiving the chemotherapy described above will have surgery to remove all or part of the breast that has cancer. If there are signs that the lymph nodes in the armpit (axilla) contain cancer, these lymph nodes will also be removed.

After chemotherapy and surgery, or after completion of chemotherapy (patients who had surgery done first), participants may then receive radiation treatment to the breast area and armpit once a day (Monday through Friday) for 5-6 weeks.

After the study, participants will return for checkups every 3-4 months during Years 1 and 2, every 6 months during years 3 and 4 and yearly after that. During the check-ups participants will talk with and be examined by their physician. Once a year, patients will have yearly mammograms (as needed), chest-x rays, and blood tests.

This is an investigational study. All of the drugs in this study are approved by the FDA for treatment of breast cancer. A total of 930 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologic confirmation of invasive, but non-inflammatory carcinoma of the breast.
2. Stage I (T1N0) are not eligible for the neo-adjuvant portion of the protocol.
3. High-risk patients (patients with any of the following: high proliferation rate - Ki67 >35% or poorly differentiated tumors (black's modified grade 3); ER/PR negative; lymphovascular invasion) with stage I disease are eligible for adjuvant therapy.
4. Patients with pure mucinous carcinomas, tubular carcinomas or pure medullary carcinomas are eligible if the patient's tumor is larger than 3 cm in size or if the patient has tumor involvement of the lymph nodes (>2mm).
5. Patients with bilateral breast cancers are eligible.
6. Patients with pN2a (metastasis in four to nine axillary lymph nodes) are eligible as are patients with pN3a (ten or more axillary lymph nodes). Patients with infraclavicular lymph node involvement are NOT eligible.
7. Patients must have clinically measurable disease to be treated in the neoadjuvant setting. This includes patients with a non-palpable primary who have histologically proven lymph node (LN) involvement that is clinically palpable and measurable by ultrasound
8. Histologic confirmation of invasive tumor will be done by core needle biopsy for patients with intact primary tumors. If patients have undergone adequate core biopsy prior to evaluation at MDACC, repeat core biopsy is optional.
9. Patients must sign an informed consent indicating that they are aware of the investigational nature of the study, in keeping with institutional policy.
10. Patients with a prior history of breast cancer are eligible if the current primary breast cancer is of a higher stage than the original breast cancer and the patient has not received any of the current study medications including past doxorubicin.
11. Patients should have adequate bone marrow function, as defined by peripheral granulocyte count of > 1,500/mm3, and platelet count > 100,000/mm3. Patients must have adequate liver function with a bilirubin within normal laboratory values. Transaminases (SGPT) may be up to 2.5x upper limit of normal (ULN) if alkaline phosphatase is < ULN or alkaline phosphatase may be up to 4 x ULN if transaminases are < ULN.
12. In addition, patients should have adequate renal function, defined as a serum creatinine < 2.5 mg% and/or creatinine clearance greater than 51 ml/min as calculated by Cockcroft and Gault Equation: Cockcroft and Gault Equation: Creatinine clearance for males = {(140 - age [yrs])(body weight [kg])}/{(72) (serum creatinine [mg/dL])}. Creatinine clearance for females = 0.85 x male value
13. Patients who had surgical therapy prior to referral will be eligible for randomization to systemic chemotherapy administered in the adjuvant setting.
14. Patients who have overexpression of the her-2/neu oncogene are eligible for the study.

Exclusion Criteria:

1. Patients with N2 (clinical staging) or N3 (clinical staging) nodal disease, inflammatory breast cancer, or metastatic disease are not eligible. This includes patients with infraclavicular and/or supraclavicular lymph node involvement. Patients with pN2a (metastasis in four to nine axillary lymph nodes) are eligible.
2. Patients with pN2b (metastasis in clinically apparent internal mammary lymph nodes in the absence of axillary lymph node metastasis) are not eligible. Patients with T4 lesions in the neoadjuvant setting are not eligible. Patients with limited T4 lesions in the adjuvant setting (for example, focal extension into the skin with negative margins) are eligible.
3. Severe hypersensitivity reactions to agents formulated in either cremophor or polysorbate 80 must be excluded. Patients with hypersensitivity reactions to any of the study medications must be excluded.
4. Those patients with history of other malignancies will be excluded, except non-melanoma skin cancer and non-invasive cervical cancer.
5. Patients with uncompensated congestive heart failure are not eligible. Patients with myocardial infarction within the past 12 months are ineligible.
6. Patients who are pregnant or lactating are not eligible. Women of childbearing potential must have a negative pregnancy test prior to initiation of chemotherapy. Women of childbearing potential who will not use a reliable and appropriate contraceptive method during the study are not eligible.
7. Patients who have had an organ allograft are ineligible.
8. Patients with serious concurrent infections are ineligible.
9. Sexually active male patients unwilling to practice contraception during the study are ineligible.
10. Patients with pre-existing peripheral neuropathy > grade 1.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 603 (Actual)
Dates: Start 2002-11; Primary Completion 2008-07 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aman U. Buzdar, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Hoon SN, Lau PK, White AM, Bulsara MK, Banks PD, Redfern AD. Capecitabine for hormone receptor-positive versus hormone receptor-negative breast cancer. Cochrane Database Syst Rev. 2021 May 26;5(5):CD011220. doi: 10.1002/14651858.CD011220.pub2. PMID 34037241
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period from November 20, 2002 to July 2, 2008. All recruitment done at UT MD Anderson Cancer Center.
Pre-assignment Details: Planned accrual was 930 participants, only 601 were found eligible.
Groups:
- Weekly Paclitaxel (WP): Weekly Paclitaxel for 12 weeks followed by Fluorouracil + Epirubicin + Cyclophosphamide (FEC) every 3 weeks for 4 cycles
- Docetaxel and Capecitabine (DX): Docetaxel + Capecitabine days 1-14 every 3 weeks for 4 cycles followed by FEC for 4 cycles.
Period: Overall Study
Arm/Group | Weekly Paclitaxel (WP) | Docetaxel and Capecitabine (DX)
Started | 302 | 301
Completed | 301 | 300
Not Completed | 1 | 1
Not completed — not eligible not invasive | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Weekly Paclitaxel (WP) | Docetaxel and Capecitabine (DX) | Total
Number analyzed (Participants) | 302 | 301 | 603
Age Continuous [Median (Full Range); unit: years] | 50 [42 to 57] | 50 [42 to 57] | 50 [42 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 302 | 301 | 603
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 302 | 301 | 603

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Reoccurrence
Description: Percentage of participants where number with local recurrence, distant metastasis, or death of any cause at 50 months is divided by total number of participants and used as primary efficacy end point to compare paclitaxel to combination docetaxel and capecitabine in breast cancer treatment for preventing recurrence (return of cancer).
Time Frame: Median of 50 months
Population: (WP Arm):301 included in the intent to treat analysis and 297 included in the safety analysis.
  (DX Arm):300 included in the intent to treat analysis and 292 included in the safety analysis.
Measure: Log Mean (95% Confidence Interval); unit: participants
Arm/Group | Weekly Paclitaxel (WP) | Docetaxel and Capecitabine (DX)
Number analyzed (Participants) | 301 | 300
participants | 90.7 [86.4 to 93.7] | 87.5 [82.7 to 91.1]

2. Secondary Outcome: Proportion of Participants With Pathological Complete Response
Description: Safety of 2 Different Treatments determined by proportion of participants who achieved pathological complete response (pCR) between two different treatments; where pCR was defined as no histopathologic evidence of any residual invasive cancer cells in the breast and axillary lymph nodes.
Time Frame: 7 Years
Reporting Status: Not Posted
Measure: Log Mean (95% Confidence Interval); unit: participants

3. Secondary Outcome: Treatment Effectiveness at Eradicating Tumor in the Breast and Lymph Nodes
Description: Effectiveness defined as proportion of patients who were able to have breast conserving surgery (BCS) after preoperative therapy compared to total number of participants.
Time Frame: 7 years
Reporting Status: Not Posted
Measure: Number; unit: participants

ADVERSE EVENTS:
Time Frame: 8 years and 5 months
Arm/Group | Weekly Paclitaxel (WP) | Docetaxel and Capecitabine (DX)
Serious Adverse Events (participants affected / at risk) | 81/301 | 293/300
Other Adverse Events (participants affected / at risk) | 297/301 | 293/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Weekly Paclitaxel (WP) (N=301) | Docetaxel and Capecitabine (DX) (N=300)
Nausea (Gastrointestinal disorders) | 5/297 (5) | 12/293 (12)
Vomiting (Gastrointestinal disorders) | 0/297 (0) | 5/293 (5)
Stomatitis (Infections and infestations) | 0/297 (0) | 5/293 (5)
Diarrhea (Gastrointestinal disorders) | 12/297 (12) | 17/293 (17)
Fatigue (General disorders) | 25/297 (25) | 66/293 (66)
Constipation (Gastrointestinal disorders) | 2/297 (2) | 6/293 (6)
Peripheral Neurotoxicity (Nervous system disorders) | 7/297 (7) | 14/293 (14)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0/297 (0) | 3/293 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 19/297 (19) | 32/293 (32)
Neutropenia (Blood and lymphatic system disorders) | 2/297 (2) | 45/293 (45)
Neutropenic Infection (Infections and infestations) | 2/297 (2) | 20/293 (20)
Neutropenic Fever (Infections and infestations) | 0/297 (0) | 13/293 (13)
Alopecia (General disorders) | 0/297 (0) | 0/293 (0)
Skin rash (Skin and subcutaneous tissue disorders) | 3/297 (3) | 1/293 (1)
Hand foot syndrome (Skin and subcutaneous tissue disorders) | 1/297 (1) | 54/293 (54)
Allergic reaction (Immune system disorders) | 2/297 (2) | 4/293 (4)
Fluid retention (Cardiac disorders) | 1/297 (1) | 0/293 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Weekly Paclitaxel (WP) (N=301) | Docetaxel and Capecitabine (DX) (N=300)
Nausea (Gastrointestinal disorders) | 64/297 (64) | 131/293 (131)
Vomiting (Gastrointestinal disorders) | 24/297 (24) | 41/293 (41)
Stomatitis (Gastrointestinal disorders) | 31/297 (31) | 118/293 (118)
Diarrhea (Gastrointestinal disorders) | 55/297 (55) | 85/293 (85)
fatigue (General disorders) | 146/297 (146) | 169/293 (169)
Constipation (Gastrointestinal disorders) | 27/297 (27) | 50/293 (50)
Peripheral Neurotoxicity (Nervous system disorders) | 68/297 (68) | 64/293 (64)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10/297 (10) | 20/293 (20)
Myalgias (Musculoskeletal and connective tissue disorders) | 109/297 (109) | 137/293 (137)
Neutropenia (Blood and lymphatic system disorders) | 30/297 (30) | 9/293 (9)
Neutropenic Infection (Blood and lymphatic system disorders) | 0/297 (0) | 0/293 (0)
Neutropenic Fever (Infections and infestations) | 0/297 (0) | 0/293 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 239/297 (239) | 266/293 (266)
Skin rash (Skin and subcutaneous tissue disorders) | 77/297 (77) | 43/293 (43)
Hand Foot Syndrome (Skin and subcutaneous tissue disorders) | 5/297 (5) | 72/293 (72)
Allergic reaction (Immune system disorders) | 4/297 (4) | 6/293 (6)
Fluid Retention (Blood and lymphatic system disorders) | 3/297 (3) | 8/293 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No